CLINICAL TRIAL: NCT06402747
Title: Comparing Clopidogrel and Cilostazol in Type 2 Diabetes Patients With Carotid Atherosclerosis
Brief Title: Clopidogrel Versus Cilostazol on Vessels
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-2401-877-002
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopidogrel (Experimental): Clopidogrel 75mg once daily
  Interventions: Drug: Clopidogrel
- Cilostazol (Active Comparator): Cilostazol 200mg per day
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75mg once daily
  Other Names: Platless Tab.
  Arms: Clopidogrel
Drug: Cilostazol — Cilostazol 200mg per day
  Other Names: Cilostan CR Tab. 200mg
  Arms: Cilostazol

SUMMARY:
Diabetes is an increasing cause of atherosclerotic and cardiovascular illnesses in South Korea. The clinical application of ultrasound for measuring carotid intima-media thickness, which helps in early detection and surveillance of atherosclerosis, is advancing. Due to lifestyle changes and an aging population, Koreans, especially diabetics, are developing more vascular diseases and are at higher risk for peripheral vascular disorders. Diabetics with lower limb peripheral artery disease require effective therapy to avoid major complications and a reduced quality of life. Although licensed for symptom control, Clopidogrel and Cilostazol have not yet been established for primary prevention of cardiovascular risks. These medications will be evaluated for their potential as primary preventive agents against cardiovascular disease in type 2 diabetes patients. The goal of this research is to investigate the efficacy of Cilostazol and Clopidogrel in inhibiting the progression of carotid atherosclerosis and to evaluate their influence on hemorheological changes in individuals with Type 2 diabetes. The goal of this research is to investigate the efficacy of Cilostazol and Clopidogrel in inhibiting the progression of carotid atherosclerosis and evaluating their influence on alterations in blood flow among individuals with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes aged 19 and older
* Individuals with a carotid ultrasound cIMT (carotid intima-media thickness) of 1.0mm or more
* Those who have not changed their combination therapy medications (including oral hypoglycemics, antihypertensives, and lipid-lowering drugs) in the last three months
* Individuals with an HbA1c level of 10% or less
* Those who have voluntarily signed the written consent form and agreed to participate in the study

Exclusion Criteria:

* Individuals currently using antithrombotic or anticoagulant medications other than aspirin
* Individuals with bleeding or conditions that may increase the risk of bleeding, such as:

  * Hemophilia, capillary fragility, intracranial hemorrhage, upper gastrointestinal bleeding, urinary bleeding, hemoptysis, vitreous hemorrhage, etc
  * Active peptic ulcer, hemorrhagic stroke within the last 6 months, surgical operations within the last 3 months, proliferative diabetic retinopathy, uncontrolled hypertension
* Patients who have had cerebrovascular or cardiovascular complications within the past 6 months (including stroke, transient ischemic attacks, myocardial infarction, unstable angina, coronary artery bypass graft, or percutaneous coronary intervention)
* Patients with severe renal or hepatic diseases
* Patients with congestive heart failure
* Individuals with a history of hypersensitivity to the drug or its components
* Pregnant women or women who may be pregnant
* Women who are breastfeeding or plan to breastfeed during the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of carotid intima-media thickness | 52 weeks
  mm

SECONDARY OUTCOMES:
Changes of circulation | 52 weeks
  measured by ankle brachial index and laser doppler
Changes of HbA1c | 26 and 52 weeks
Changes of glucose | 26 and 52 weeks
  mg/dL
Changes of body weight | 26 and 52 weeks
  kg
Changes of whole body fat | 26 and 52 weeks
  measured by bioelectrical impedance analysis
Changes of blood pressures | 26 and 52 weeks
  systolic, diastolic (mmHg)
Changes of lipids | 26 and 52 weeks
  total cholesterol, triglycerides, LDLc, HDLc (mg/dL)
Changes of peripheral pain or ischemic symptoms | 26 and 52 weeks
  measured by questionnaires (visual analogue scale: 100)
Changes of laboratory values related to blood clot | 26 and 52 weeks
  prothrombin time, activated partial thromboplastin time

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD. Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No